CLINICAL TRIAL: NCT01393665
Title: Multicenter, Randomized, Placebo-Controlled, Double-blind Phase 2 Study to Evaluate the Short-term Efficacy, Safety and Tolerance and to Find an Optimal Dosage of the PENNEL Capsule for the Patients With Chronic Liver Disease
Brief Title: Study to Evaluate Efficacy, Safety and Tolerability of PENNEL Capsule in the Patients With Chronic Liver Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaKing (Industry)
Responsible Party: R&D department, CR team
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PMK-PENNEL 2
Record Dates: First submitted 2011-07-03; First posted 2011-07-13 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- PENNEL capsule (Experimental): 1cap or 2cap T.I.D
  Interventions: Drug: PENNEL capsule

INTERVENTIONS:
Drug: PENNEL capsule — hard capsule DDB 25mg & GO 50mg in cap .......... 1 capsule
  1 or 2 capsule, T.I.D
  Arms: PENNEL capsule
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The test agent in this study is a product of biphenylmethyl dicarboxylate (BDD) with garlic oil. The two components were confirmed to have complementary effects because of different operational mechanism in animal experiments, and were examined on humans in this study. Both BDD and garlic oil are expected to show better protection and treatment on hepatotoxicity caused by toxic substances, and the purpose of this study is to confirm efficacy of and safety on human body of the agent and to determine its optimal dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic liver disease.
* Patients over 20, under 65 years of age.
* Patients with abnormal transaminase levels.

Exclusion Criteria:

* Pregnant and lactating women.
* Patients who have any history of esophageal bleeding, hepatic encephalopathy, ascites.
* Diabetes, thyroid dysfunction, fatty liver, liver cancer patients.
* Toxic hepatitis, alcoholic hepatitis.
* Total bilirubin value more than 3.0 mg/dl.
* Albumin value less than 3.0 g/dl.
* Patients who participating in other study about drug.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 1996-12; Primary Completion 1997-05 (Actual); Study Completion 1997-10 (Actual)

PRIMARY OUTCOMES:
ALT (Alanine Aminotransferase) | 6 week
  To evaluate the efficacy of the PENNEL capsule on change ALT from baseline to 6 weeks (Change from Baseline in Alanine Aminotransferase at 6 weeks)
  The measurements were conducted five times, including ① before administration, ② the 1st week of administration, ③ the 3rd week of administration, ④ the 6th week of administration, and ⑤ the 1st week after the six-week administration.

SECONDARY OUTCOMES:
AST (Aspartate Aminotransferase) | 6 weeks
  To evaluate the efficacy of the PENNEL capsule on change AST from baseline to 6 weeks (Change from Baseline in Aspartate Aminotransferase at 6 weeks)
  The measurements were conducted five times, including ① before administration, ② the 1st week of administration, ③ the 3rd week of administration, ④ the 6th week of administration, and ⑤ the 1st week after the six-week administration.
g-GT (γ-glutamyl transpeptidase) | 6 weeks
  To evaluate the efficacy of the PENNEL capsule on change g-GT from baseline to 6 weeks (Change from Baseline in γ-glutamyl transpeptidase at 6 weeks)
  The measurements were conducted five times, including ① before administration, ② the 1st week of administration, ③ the 3rd week of administration, ④ the 6th week of administration, and ⑤ the 1st week after the six-week administration.
Total bilirubin | 6 weeks
  To evaluate the efficacy of the PENNEL capsule on change Total bilirubin from baseline to 6 weeks (Change from Baseline in Total bilirubin at 6 weeks)
  The measurements were conducted five times, including ① before administration, ② the 1st week of administration, ③ the 3rd week of administration, ④ the 6th week of administration, and ⑤ the 1st week after the six-week administration.

CONTACTS AND LOCATIONS:
Overall Officials: Minho Lee, MD.PhD, Principal Investigator — Hanyang University
Locations (2):
- South Korea (2):
  - Korea Cancer Center Hospital, Seoul, Nowon-gu
  - Hanyang University Hospital, Seoul, Seongdong-gu

REFERENCES:
- [Derived] Lee MH, Kim YM, Kim SG. Efficacy and tolerability of diphenyl-dimethyl-dicarboxylate plus garlic oil in patients with chronic hepatitis. Int J Clin Pharmacol Ther. 2012 Nov;50(11):778-86. doi: 10.5414/CP201746. PMID 22943930